CLINICAL TRIAL: NCT02334579
Title: Function-Preserving Stereotactic Body Radiotherapy for Clinical State I-III Prostate Cancer
Brief Title: Stereotactic Body Radiotherapy for Stage I-III Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR 5642
Record Dates: First submitted 2014-12-04; First posted 2015-01-08 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer; Prostatic Cancer; Prostate Neoplasms; Prostatic Neoplasms; Cancer of the Prostate
Keywords: Radiation; Stereotactic Radiosurgery; Radiotherapy; Prostate Tumor; Prostate Surgery; CyberKnife
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyberKnife Stereotactic Radiosurgery (Experimental): This treatment concentrates large doses of radiation onto the tumor so that injury from radiation to the nearby normal tissue will be minimal. CyberKnife Stereotactic Radiosurgery is not investigational and is considered standard of care.
  Interventions: Radiation: CyberKnife Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: CyberKnife Stereotactic Radiosurgery — Five treatments given over about one week.

SUMMARY:
The purpose of this study is to find out the effects (good and bad) of highly focused radiation on you and your prostate cancer. The purpose of this evaluation is to see if this treatment causes fewer side effects that other standard treatment approaches, and to evaluate the effect of this treatment on your prostate tumor and your quality of life over time.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate adenocarcinoma
* Clinical stage T1a-T3, N0-Nx, M0-Mx
* Patients belonging in one of the following risk groups: (1) LOW RISK: CS T1a-T2a, Gleason 2-6, PSA<10, Nx-0, Mx-0; (2) INTERMEDIATE RISK: CS T2b, Gleason ≤7, PSA<20, Nx-0, Mx-0, or CS T1a-T2b, Gleason 2-6, PSA≥10 & <20, Nx-0, Mx-0, or CS T1a-T2b, Gleason 7, PSA≤20, Nx-0, Mx-0; or (3) HIGH RISK: CS T2c-T3, any Gleason, any PSA, or CS T1-3, Gleason ≥8 and/or PSA≥20
* Karnofsky performance status 70-100
* Hormone therapy: includes LHRH agonists (e.g. leuprolide, goserelin, triptorelin), antagonists (e.g. degarelix), peripheral blockers (e.g. flutamide, bicalutamide, nilutamide), estrogens (e.g. DES) and bilateral orchiectomy
* Low and Intermediate risk groups: no hormone ablation for two months prior to enrollment, or during treatment
* High risk group: three hormone therapy regimens are allowed
* 5-alpha reductase inhibitors (e.g., finasteride or dutasteride) are allowed

Exclusion Criteria:

* Prior prostatectomy or cryotherapy of the prostate
* Prior high-dose radiotherapy to the prostate or lower pelvis
* Implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2014-12; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life outcomes (low- and intermediate-risk prostate cancer groups) | 8 years
  In the low- and intermediate-risk prostate cancer groups, to determine whether study treatment improves patient-reported quality of life outcomes compared to the approach used in a previous multi-center cyberknife stereotactic radiosurgery trial.
Rates of acute and late grade 3-5 gastrointestinal and genitourinary toxicities (high-risk group) | 8 years
  In the high-risk group, to estimate rates of acute and late grade 3-5 gastrointestinal and genitourinary toxicities following cyberknife stereotactic radiosurgery.

SECONDARY OUTCOMES:
Rates of toxicities related to treatment | 5 years
  After five years following cyberknife stereotactic radiosurgery, estimate rates of toxicities related to treatment.
Disease free survival | 5 years
  Measure disease free survival after five years following cyberknife stereotactic radiosurgery.
Overall survival | 5 years
  Measure overall survival after five years following cyberknife stereotactic radiosurgery.

OTHER OUTCOMES:
Quality of life | 5 years
  Measure quality of life after five years following cyberknife stereotactic radiosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Meier, MD, Principal Investigator — Swedish Medical Center Radiosurgery Center
Locations (1):
- Swedish Medical Center Radiosurgery Center, Seattle, Washington, United States

REFERENCES:
- See also: Swedish Medical Center Radiosurgery Center — http://www.swedish.org/services/radiosurgery-center